CLINICAL TRIAL: NCT01725893
Title: Percutaneous Tenotomy of the Toe Flexor Tendon is a Simple and Efficient Method in Treating Checkrein Deformity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, National Taiwan University Hospital (NTUH) Research Ethics Committee (REC), National Taiwan University Hospital
Other Study IDs: 201202038RIC
Record Dates: First submitted 2012-09-25; First posted 2012-11-14 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Claw Toe
Keywords: Claw Toe
MeSH Terms: conditions — Hammer Toe Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Checkrein deformity represents a dynamic claw toe deformity. Surgical intervention is the treatment of choice and many methods have been proposed. The purpose of this study is to evaluate the outcomes and complications of percutaneous segmental tenotomy of the toe flexor tendons.

DETAILED DESCRIPTION:
The investigators reviewed fourteen patients with checkrein deformity who underwent surgery in our hospital between 1993 and 2010. Five patients received FHL and flexor digitorum longus (FDL) tenolysis at the musculotendinous junction; among them, two also underwent Z-plasty lengthening of the FHL tendon. Nine patients underwent percutaneous segmental toe flexor tenotomy. The Hallux Metatarsophalangeal- Interphalangeal Scale (Hallux MTP-IP scale) and Foot and Ankle Outcome Score (FAOS), English version LK1.0 self-explanatory questionnaire were used to evaluate the functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with checkrein deformity who underwent surgery in our hospital between 1993 and 2010.

Exclusion Criteria:

* Patients who had static or rigid claw toe deformity
* Patients who had claw toe deformity secondary to neuromuscular disease

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There were fourteen patients with checkrein deformity who underwent surgery in our hospital between 1993 and 2010.
Sampling Method: Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-01 (Estimated); Study Completion 2013-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hong-Nerng Ho, Professor, Study Chair — National Taiwan University Hospital (NTUH) Research Ethics Committee (REC)
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Result] Lee HS, Kim JS, Park SS, Lee DH, Park JM, Wapner KL. Treatment of checkrein deformity of the hallux. J Bone Joint Surg Br. 2008 Aug;90(8):1055-8. doi: 10.1302/0301-620X.90B8.20563. PMID 18669962